CLINICAL TRIAL: NCT01412476
Title: Coenzyme Q10 and Vitamin A, C, E in Relation to the Oxidative Stress, Antioxidant Enzyme Activity and Inflammation in Subjects With Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Ping-Ting Lin, Chung Shan Medical University
Other Study IDs: CS09155
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case group: Subjects with metabolic syndrome
- control group: Healthy individuals

SUMMARY:
Metabolic syndrome (MS) is a significant risk factor of cardiovascular disease. However, the relationships between coenzyme Q10, antioxidant vitamins (Vitamin A, C, E) and the prevention of the risk of MS are still inconsistent. The purposes of this study are going to investigate the relation of coenzyme Q10, antioxidant vitamins concentration with the blood lipid levels, the markers of lipid peroxidation (TBARS), antioxidant enzymes activities (catalase, glutathione peroxidase and superoxide dismutase), and the inflammatory markers (hs-CRP,IL-6 and adiponectin). The investigators will recruit MS patients (case group, n = 100) and age-gender matched healthy subjects from previous study(n = 105) as a control group . The inclusion criteria of MS are according to the Bureau of Health Promotion, Department of Health in Taiwan (2007).Hopefully, the results of this study could provide the information to what has been know in MS subjects. The investigators expect coenzyme Q10 or antioxidant vitamins could be a preventive supplement to reduce the risk of MS.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome
* Healthy individuals with normal blood biochemical values.

Exclusion Criteria:

* Age < 18y
* Antioxidant vitamins supplements use
* Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators recruited MS patients (case group, n = 100). The inclusion criteria of MS are according to the Bureau of Health Promotion, Department of Health in Taiwan (2007). The health subject were recrited from previous study (n = 105).
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2010-08; Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ting Lin, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Ping-Ting Lin, Taichung, Taiwan